CLINICAL TRIAL: NCT00951197
Title: Estimation of Microstructure Alteration by MRI in Dementia Among Elderly Subjects Retired From Agricultural Profession and Living in Rural Area in Gironde - Participants From the AMI Cohort.
Brief Title: Evaluation of Alteration by Magnetic Resonance Imaging (MRI) in Dementia Among Elderly Subjects
Acronym: AMIMAGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2008/13
Record Dates: First submitted 2009-04-22; First posted 2009-08-04 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Dementia; Alzheimer Disease
Keywords: dementia; Alzheimer's Disease; diagnostic; biomarkers; neuroimaging; PET; MRI; mild cognitive impairment
MeSH Terms: conditions — Dementia; Alzheimer Disease; Disease; Cognitive Dysfunction | interventions — Neuroimaging

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- elderly subjects retired from agriculture
  Interventions: Other: Neuroimaging

INTERVENTIONS:
Other: Neuroimaging — Three successive MRI acquisitions to measure FA, MTR and T2 parameters.

SUMMARY:
Capturing the earliest stages of Dementia especially Alzheimer's Disease (AD) is a great challenge. Until now the NINCDS-ADRDA and the DSM criteria for AD were largely used as diagnostic standards in research. However, the research on AD progresses and some biomarkers have been recently suggested to improve the diagnostic criteria of AD, such as cerebrospinal fluid markers, neuroimaging with Positon Emission Tomography (PET) or Magnetic Resonance Imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* participate in the AMI cohort
* be aged 65 and older
* be retired from agricultural profession
* live in rural area in Gironde

Exclusion Criteria:

* contraindication of MRI
* left-handed
* severe dementia
* Parkinson's disease
* poor health incompatible with the transport to neuroimaging service
* to be left handed

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: population retired from agricultural profession and living in rural area in Gironde
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
FA (Fractional Anisotropy), MTR (magnetization transfer ratio) and T2 (Transverse relaxation time) measures in patients with dementia compared to controls, in left and right hippocampus, and posterior cingulum | day 0

SECONDARY OUTCOMES:
FA, MTR and T2 measures in subjects with mild cognitive impairment no dementia | day 0
Performances in the 7 neuropsychological tests available in the AMI cohort | day 0
FA measures for the connexion Hippocampus-cingulum posterior | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Michèle ALLARD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Groupe Hospitalier Pellegrin - C.H.U. de Bordeaux, Bordeaux, France